CLINICAL TRIAL: NCT00078195
Title: Efficacy and Safety Evaluation of Allergen Immunotherapy Co-Administered With Omalizumab, an Anti-IgE Monoclonal Antibody (ITN019AD)
Brief Title: Omalizumab (Xolair) and Allergy Shots For the Treatment of Seasonal Allergies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN019AD
Record Dates: First submitted 2004-02-19; First posted 2004-02-20 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hay Fever; Hypersensitivity; Allergy; Rhinitis
Keywords: Ragweed; Immunotherapy; Rush Immunotherapy; RIT; Hayfever; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Rhinitis | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Omalizumab pre-treatment, ragweed RIT, omalizumab + ragweed IT (Experimental): Participants are pre-treated with omalizumab followed by ragweed rush immunotherapy (RIT) followed by dual therapy with omalizumab plus ragweed immunotherapy (IT).
  Interventions: Biological: omalizumab; Biological: Ragweed rush immunotherapy (RIT); Biological: Ragweed immunotherapy (IT)
- Omalizumab pre-treatment, omalizumab (Experimental): Participants are pre-treated with omalizumab followed by placebo rush immunotherapy (RIT), followed by dual therapy with Omalizumab plus placebo immunotherapy (IT).
  Interventions: Biological: omalizumab; Biological: Placebo rush immunotherapy (RIT); Biological: Placebo immunotherapy (IT)
- Ragweed RIT, ragweed IT (Active Comparator): Participants are pre-treated with placebo omalizumab followed by ragweed rush immunotherapy (RIT), followed by dual therapy with placebo omalizumab plus ragweed immunotherapy (IT).
  Interventions: Biological: Placebo omalizumab; Biological: Ragweed rush immunotherapy (RIT); Biological: Ragweed immunotherapy (IT)
- Placebo (Placebo Comparator): Participants are pre-treated with placebo omalizumab followed by placebo rush immunotherapy (RIT), followed by dual therapy with placebo omalizumab plus placebo immunotherapy (IT).
  Interventions: Biological: Placebo omalizumab; Biological: Placebo rush immunotherapy (RIT); Biological: Placebo immunotherapy (IT)

INTERVENTIONS:
Biological: omalizumab — A minimum equivalent dose of 0.016 mg/kg/IgE (IU/mL) every 4 weeks will be administered. Omalizumab is administered in two separate phases. In the pre-treatment period omalizumab will be administered to condition the participants to an immune tolerance state. Omalizumab will be also administered after RIT and during the maintenance immunotherapy phase.
  Other Names: Xolair™; anti-Immunoglobulin E (IgE)
  Arms: Omalizumab pre-treatment, omalizumab; Omalizumab pre-treatment, ragweed RIT, omalizumab + ragweed IT
Biological: Placebo omalizumab — The placebo for omalizumab will contain the excipients and diluents of the omalizumab.
  Arms: Placebo; Ragweed RIT, ragweed IT
Biological: Ragweed rush immunotherapy (RIT) — RIT will consist of a series of injections containing ragweed extract. The series of injections will have progressively greater amounts of ragweed extract: starting from the 1:1000 dilution of the maintenance vial and progressing to the 0.3 mL of 1:10 dilution of the maintenance vial or the maximally tolerated amount.
  Arms: Omalizumab pre-treatment, ragweed RIT, omalizumab + ragweed IT; Ragweed RIT, ragweed IT
Biological: Placebo rush immunotherapy (RIT) — The placebo for rush immunotherapy will contain the diluents and histamine.
  Arms: Omalizumab pre-treatment, omalizumab; Placebo
Biological: Ragweed immunotherapy (IT) — Participants will receive weekly maintenance IT dosing for a total of 12 weeks.
  Arms: Omalizumab pre-treatment, ragweed RIT, omalizumab + ragweed IT; Ragweed RIT, ragweed IT
Biological: Placebo immunotherapy (IT) — The placebo for immunotherapy will contain the diluents and histamine.
  Arms: Omalizumab pre-treatment, omalizumab; Placebo

SUMMARY:
A series of allergy shots may reduce symptoms of seasonal ragweed allergies. This study will determine whether taking a drug called omalizumab (also known as Xolair) before getting the allergy shots is more effective than allergy shots alone or other treatments, such as prescription antihistamines.

DETAILED DESCRIPTION:
Allergic rhinitis affects 20 to 40 million Americans annually. Allergy symptoms, which can range from mild to seriously debilitating, may affect quality of life. Left untreated, allergic rhinitis can exacerbate or trigger more serious conditions, such as asthma and sinus inflammation.

Individuals with allergies react to harmless particles such as dust or pollen. Proteins in the blood called IgE antibodies treat the harmless particles as invaders and trigger an immune system response. The immune response results in harmful inflammation of healthy tissues. In ragweed allergy, inflammation occurs in the airways and causes familiar allergy symptoms like sneezing, coughing, and general discomfort.

Omalizumab is an investigational drug that has been shown to block the effects of IgE antibodies. The blocking effect of omalizumab is temporary, but giving the drug to people before their regular allergy shots may make the shots more effective.

Participants in this study will be randomly assigned to receive injections of omalizumab or a placebo before an accelerated course of allergy shots (given over 12 weeks). The participants will return for follow-up for up to one year, and they may have as many as 27 study visits.

ELIGIBILITY:
Inclusion Criteria

* Able to comprehend and grant a witnessed, written informed consent prior to any study procedures.
* Female participants of child bearing age must have a negative urine pregnancy test at Screening Visit and subsequent visits. In addition, female participants must be using a medically acceptable form of birth control.
* History of seasonal allergic rhinitis for at least 2 years with symptoms during the ragweed pollen season requiring pharmacotherapy.
* A positive skin test by prick method to ragweed pollen at the Screening Visit. A positive skin prick test will be defined as a ragweed pollen-induced wheal greater than 3 mm larger in diameter than diluent control (measurements will be made 15-20 minutes after application).
* Must be capable of faithfully completing the diary and of attending regularly scheduled study visits.
* Must intend to remain in the ragweed pollen area during the entire ragweed season.
* Willing to avoid prohibited medications for the periods indicated in the protocol.
* Participants must meet pretrial eligibility requirements for trial enrollment (acceptable medical history, physical examination results, normal electrocardiogram and acceptable laboratory test results).
* Participants must have a baseline serum Immunoglobulin E (IgE) level greater than 10 and less than 700 IU/mL.

Exclusion Criteria

* weigh less than 30 kg or more than 120 kg.
* pregnant or lactating.
* history of severe anaphylactoid (non-IgE mediated) or anaphylactic reactions).
* history of immunotherapy within the past 10 years, if received one full year of immunotherapy, or within the past 5 years if received less than one year of immunotherapy.
* known hypersensitivity to trial rescue medication (fexofenadine HCl).
* taking beta-adrenergic antagonists in any form.
* taking allergic ophthalmologic medication.
* clinically significant perennial rhinitis that would interfere in assessment of ragweed-induced seasonal allergic rhinitis symptoms.
* Presence of a severely deviated nasal septum, septal perforation, structural nasal defect or large nasal polyps causing obstruction.
* History of an upper respiratory or sinus infection requiring treatment with an antibiotic within 2 weeks prior to Screening Visit.
* Documented evidence of acute or significant chronic sinusitis, as determined by the Investigator.
* Asthma (either history of, abnormal spirometry, [forced expiratory volume in 1 second (FEV1) less than 80% predicted] or use of asthma medications).
* Chronic or intermittent use of inhaled, oral, intra-muscular, or intra-venous corticosteroids; or chronic or intermittent use of topical corticosteroids within 4 weeks of Visit Screening Visit.
* Chronic use of medications (e.g., tricyclic antidepressants) that would affect assessment of the effectiveness of the study medication.
* Rhinitis medicamentosa.
* History or presence of significant renal, hepatic, neurologic, cardiovascular, hematologic, metabolic, cerebrovascular, respiratory, gastrointestinal or other significant medical condition including, autoimmune or collagen vascular disorders, aside from organ-specific autoimmune disease limited to the thyroid that in the Investigator's opinion could interfere with the study or require medical treatment that would interfere with the study.
* History of cancer other than basal cell carcinoma of the skin.
* History within the past year of excessive alcohol intake or drug addiction.
* Current smokers, greater than 10 pack year history, or participants who quit smoking less than one year prior to Screening.
* Use of any prohibited concomitant medications during the washout period (i.e., before screening) and throughout the study period.
* Participants currently undergoing immunotherapy.
* Participants with clinically significant abnormality on 12-lead Electrocardiogram (ECG) on screening visit.
* Treatment with an experimental, non-approved drug, or investigational drug within the past 30 days.
* Participants with a history of noncompliance to medical regimens and participants who are considered potentially unreliable.
* Previous treatment with a monoclonal antibody for any reason including anti-IgE in any form (e.g., omalizumab).
* Participants with known hypersensitivity to trial drug ingredients (i.e., sucrose, histidine, polysorbate 20) or related drugs (i.e., monoclonal antibody; polyclonal gamma-globulin).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168
Dates: Start 2003-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Average daily allergy severity score | 2003 ragweed pollen season
  The average daily allergy severity score will be calculated from participants' 5 symptom scores (sneezing; rhinorrhea/runny nose; itchy nose, throat, and palate; itchy, watery eyes; and nasal congestion/stuffiness) during the ragweed pollen season. Symptom scores are recorded twice daily (AM and PM). The sum of the individual symptom scores will be averaged over AM and PM to give a daily score. Each daily score will then be averaged to obtain one measure of the average daily allergy severity score for each participant. The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.
Number of days with rescue medication (fexofenadine HCl 60 mg) use | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.
Number of rescue medication capsules used | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.
Rhinoconjunctivitis quality of life (QOL) questionnaire (RQLQ) scores | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.
Daily morning allergy symptom scores | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.
Daily nighttime allergy symptom scores during the 2003 ragweed season | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.
Individual allergy symptom scores during the 2003 ragweed season | 2003 ragweed pollen season
  The ragweed pollen season begins when the ragweed pollen counts rise to 10 ragweed pollen grains/m3/24 hours or above on two consecutive recorded days, and the ragweed pollen season ends when the ragweed pollen counts fall below 10 ragweed pollen grains/m3/24 hours on two consecutive recorded days. The ragweed pollen season is from approximately August 15, 2003 to October 1, 2003, but varies among the sites.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Casale, MD, Principal Investigator — Creighton University
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Creighton University, Omaha, Nebraska
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in: 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research data sharing portal.

REFERENCES:
- [Result] Nayak A, Casale T, Miller SD, Condemi J, McAlary M, Fowler-Taylor A, Della Cioppa G, Gupta N. Tolerability of retreatment with omalizumab, a recombinant humanized monoclonal anti-IgE antibody, during a second ragweed pollen season in patients with seasonal allergic rhinitis. Allergy Asthma Proc. 2003 Sep-Oct;24(5):323-9. PMID 14619332
- [Result] Casale TB, Busse WW, Kline JN, Ballas ZK, Moss MH, Townley RG, Mokhtarani M, Seyfert-Margolis V, Asare A, Bateman K, Deniz Y; Immune Tolerance Network Group. Omalizumab pretreatment decreases acute reactions after rush immunotherapy for ragweed-induced seasonal allergic rhinitis. J Allergy Clin Immunol. 2006 Jan;117(1):134-40. doi: 10.1016/j.jaci.2005.09.036. Epub 2005 Dec 2. PMID 16387596
- [Result] Klunker S, Saggar LR, Seyfert-Margolis V, Asare AL, Casale TB, Durham SR, Francis JN; Immune Tolerance Network Group. Combination treatment with omalizumab and rush immunotherapy for ragweed-induced allergic rhinitis: Inhibition of IgE-facilitated allergen binding. J Allergy Clin Immunol. 2007 Sep;120(3):688-95. doi: 10.1016/j.jaci.2007.05.034. Epub 2007 Jul 12. PMID 17631952
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY1 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY1 — ImmPort study identifier is SDY1
- Available data/document: Study Protocol: SDY1 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY1 — ImmPort study identifier is SDY1
- Available data/document: Study design, -summary, -files, -interventions, participant schedule of events, -demographics, et al.: SDY1 — http://www.itntrialshare.org/project/Studies/ITN019ADPUBLIC/Study%20Data/begin.view? — ImmPort study identifier is SDY1
- Available data/document: Individual Participant Data Set: CASALE ITN019AD — http://www.itntrialshare.org/project/Studies/ITN019ADPUBLIC/Study%20Data/begin.view? — TrialShare study identifier is CASALE ITN019AD
- Available data/document: Study protocol synopsis; -schedule of assessments; -data and reports; -specimens availability et al.: CASALE ITN019AD — http://www.itntrialshare.org/project/Studies/ITN019ADPUBLIC/Study%20Data/begin.view? — TrialShare study identifier is CASALE ITN019AD